CLINICAL TRIAL: NCT02668237
Title: Impact on Anti-infectious Treatments of the Early Molecular Detection Technique Coupled With Urinary Test of Infectious Agents Responsible of Community-acquired Pneumonia of Children at Pediatric Emergencies
Brief Title: Early Molecular Detection Technique Coupled With Urinary Test of Infectious Agents Responsible of Children CAP
Acronym: OptiPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1508188; 16-367 (Other: CCTIRS); 916352 (Other: CNIL); 2016-A00483-48 (Other: ANSM)
Record Dates: First submitted 2016-01-22; First posted 2016-01-29 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Community-Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The intervention for this group will be the use of a OptiPAC. A molecular technique and urinary tests will be performed to test a panel of infectious agents : the results will allow the children to benefit from an adapted treatment.
  Interventions: Other: OptiPAC
- Control Group (Active Comparator): The children will benefit from the usual care : an antibiotic prevention treatment.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: OptiPAC — Molecular and urinary tests.
  Arms: Experimental group
Other: Usual care — Antibiotics for prevention.
  Arms: Control Group

SUMMARY:
Community-Acquired Pneumonia (CAP) of children are a recurrent pathology with multiple severity scores. The etiology is never really identified, and the initial treatment is always based on probabilistic antibiotics, in the case of an bacterial infection, and by the way, potentially severe.

Molecular tests ("multiplex") allow the simultaneous detection of a huge number of pathogenic agents, virus and bacteria, are now available.

This project is based on a new strategy of diagnostic, using a multiplex PCR with quick results, coupled to an antigenic urinary test to allow a complete, quick, etiologic diagnostic as soon as children are supported in emergency.

Children are randomized in two groups during inclusions : quick diagnostic strategy versus usual practice. Analyse will be centralized on anti-infectious treatment optimization, with the aim to better treat patients, minimize the costs, and decrease selection pressure of multi-resistant bacteria.

DETAILED DESCRIPTION:
Community-Acquired Pneumonia (CAP) of children are a recurrent pathology with multiple severity scores. Almost two out of three cases identified at emergency are treated in ambulatory because patients present a reassuring clinical state. The etiology is never really identified, and the initial treatment is always based on probabilistic antibiotics re-evaluated at H48, in the case of an bacterial infection, and by the way, potentially severe. This old conception is opposed to the new discoveries, more particularly in pediatric units where strictly viral pneumonia are more important than predicted (at least 30 to 50%) that leads to an hyper prescription of antibiotics, useless.

Molecular tests ("multiplex") allow the simultaneous detection of a huge number of pathogenic agents, virus and bacteria, are now available.

Aware of the non specificity of the clinical data to guide the diagnostic, this project is based on a new strategy of diagnostic, using a multiplex PCR with quick results (less than 2 hours, for 20 pathogens, including 17 viruses) coupled to an antigenic urinary test to allow a complete, quick, etiologic diagnostic as soon as children are supported in emergency.

Children are randomized in two groups during inclusions : quick diagnostic strategy versus usual practice. Analyse will be centralized on anti-infectious treatment optimization (antibiotics and antiviruses), with the aim to better treat patients, minimize the costs, and decrease selection pressure of multi-resistant bacteria.

ELIGIBILITY:
Inclusion Criteria:

* In emergency for a Community-Acquired Pneumonia (according to the international rules based on an hyperthermia > 38,5°C associated to a radiological opacity)
* Informed Consent
* Possibility to take samples

Exclusion Criteria:

* Nosocomial pneumonia
* Pleuropneumopathy
* Pneumonia occurring in immunosuppressed and transplanted
* Patient with proven allergy to antibiotics
* Inability to perform certain microbiological samples

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Appropriate prescription of an anti-infection treatment. | Day 1
  Measure the impact on the therapeutic support of the creation of a quick, diagnostic, etiologic test of Community-Acquired Pneumonia of children (less than 3 months), supported in pediatric emergency versus usual practice. The main criterion will be the appropriate prescription of an anti-infection treatment, taking into account the microbiological results obtained a posteriori and clinical evolution. The primary outcome will be measured directly in the patients source folders.

CONTACTS AND LOCATIONS:
Overall Officials: CANTAIS Aymeric, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (11):
- France (11):
  - Chu Marseille, Marseille, La Timone
  - Chu Saint Etienne, Saint-Etienne, Saint Etienne
  - Chu Brest, Brest
  - CHU CAEN, Caen
  - Chu Estaing, Clermont-Ferrand
  - Chu Grenoble, Grenoble
  - APHP - Béclère, Paris
  - APHP - Necker, Paris
  - Chu Reims, Reims
  - Chu Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cantais A, Pillet S, Rigaill J, Angoulvant F, Gras-Le-Guen C, Cros P, Thuiller C, Molly C, Tripodi L, Desbree A, Annino N, Verhoeven P, Carricajo A, Bourlet T, Chapelle C, Claudet I, Garcin A, Izopet J, Mory O, Pozzetto B; OPTIPAC study group. Impact of respiratory pathogens detection by a rapid multiplex polymerase chain reaction assay on the management of community-acquired pneumonia for children at the paediatric emergency department. A randomized controlled trial, the Optimization of Pneumonia Acute Care (OPTIPAC) study. Clin Microbiol Infect. 2025 Jan;31(1):64-70. doi: 10.1016/j.cmi.2024.08.001. Epub 2024 Aug 5. PMID 39111697